CLINICAL TRIAL: NCT04238572
Title: Evaluation of an Immersive Audiovisual Distraction Device Impact on Peroperative Opioid Consumption. A Prospective Randomized Controlled Study
Brief Title: Evaluation of Immersive Audiovisual Distraction Impact on Peroperative Opioid Consumption.
Acronym: AmbuCineView
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-A01243-54
Record Dates: First submitted 2020-01-17; First posted 2020-01-23 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-01

CONDITIONS: Surgical Procedure, Unspecified; Analgesia; Outpatient
Keywords: Audiovisual distraction device; Peroperative opioid analgesia; Ambulatory care; Outpatient; Analgesia nociception index; Anxiety; Remifentanil; Remifentanil added to local anesthesia
MeSH Terms: conditions — Agnosia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: 200 patients will be randomized. 100 patients operated on in vitro fertilization (50 patients in intervention group, 50 patients in active comparator group) 100 patients operated on venous access port placement (50 patients in intervention group, 50 patients in active comparator group)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audiovisual distraction device (Experimental): Audiovisual distraction device, analgesia nociception index monitoring, remifentanil added to local anesthesia technique
  Interventions: Device: Audiovisual distraction device; Device: Analgesia nociception index
- Active comparator group (Active Comparator): Analgesia nociception index monitoring, remifentanil added to local anesthesia technique
  Interventions: Device: Analgesia nociception index

INTERVENTIONS:
Device: Audiovisual distraction device — Evaluate the impact of an audiovisual distraction device on the peroperative opioid consumption
  Arms: Audiovisual distraction device
Device: Analgesia nociception index — ANI (Analgesia Nociception Index) will be used for peroperative overall comfort measurement

SUMMARY:
This study evaluate the impact of an audiovisual distraction device on the peroperative opioid consumption for outpatient procedures with Remifentanil added to local anesthesia.

Half of patients will receive an audiovisual distraction device while the other half not.

DETAILED DESCRIPTION:
Early recovery for patients undergoing surgery is the key factor for an outpatient procedure.

The technique of adding remifentanil to a local anesthesia is used in 22% of the procedures realized in The CHU de Caen Outpatient unit. Decreasing opioid dose, whose side effects are numerous and widely described, as well as reducing anxiety are daily challenges to ensure comfort and successful care.

We propose a prospective, randomized, monocentric, open label study to evaluate the impact of the use of an audiovisual distraction device on the intraoperative consumption of opioids, on the patient's pain and peroperative anxiety.

ANI (Analgesia Nociception Index) will be used for peroperative overall comfort measurement. We will analyze if audiovisual distraction can integrate existing techniques such as hypnosis.

Finally, we will also assess the medico-economic impact of this technique in order to establish a benefit / cost ratio.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Signed consent
* Outpatient surgery eligibility
* Patient covered by social security

Exclusion Criteria:

* Unsigned consent
* Study participation refusal
* Deafness, blindness
* Claustrophobia
* ANI contraindication (atrial fibrillation, pace maker, severe autonomic system dysfunction)
* Contraindication or impossibility to use the audiovisual distraction device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative Remifentanil dose | 1 hour
  μg/kg/min

SECONDARY OUTCOMES:
Preoperative pain measured with a numeric pain rating scale (NRS) | 1 hour
  Numeric pain rating scale (0 = No pain to 10 = Worst pain imaginable)
Preoperative anxiety measured by the Amsterdam Preoperative Anxiety and Information Scale (APAIS) | 1 hour
  APAIS measures the need-for-information with 6 items. Each one is rated from 1 = Not at all to 5 = Extremely. There is positive and significant correlation between the ned-for-information and anxiety.
Preoperative anxiety measured by a visual analogue scale (VAS) | 1 hour
  Visual analogue scale is a 100mm horizontal line. At the left hand (0mm) the statement "not anxious at all" and at the right hand (100mm) the statement "most anxious I can imagine"
Per operative Analgesia nociception index (ANI) value | 1 hour
  From 0 = Predominant sympathetic tone, pain and anxiety to 100 = Predominant parasympathetic tone, good analgesia.
  Negative linear Relationship between analgesia nociception index and pain scores
Post operative anxiety measured by a visual analogue scale (VAS) | 1 hour
  Visual analogue scale is a 100mm horizontal line. At the left hand (0mm) the statement "not anxious at all" and at the right hand (100mm) the statement "most anxious I can imagine"
Postoperative pain measured with a numeric pain rating scale (NRS) | 1 hour
  Numeric pain rating scale (0 = No pain to 10 = Worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Clément Buléon, MD, Study Chair — Caen UH
Locations (1):
- Caen University Hospital, Caen, Calvados, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marsdin E, Noble JG, Reynard JM, Turney BW. Audiovisual distraction reduces pain perception during shockwave lithotripsy. J Endourol. 2012 May;26(5):531-4. doi: 10.1089/end.2011.0430. Epub 2012 Feb 8. PMID 22098167
- [Background] Lee DW, Chan AC, Wong SK, Fung TM, Li AC, Chan SK, Mui LM, Ng EK, Chung SC. Can visual distraction decrease the dose of patient-controlled sedation required during colonoscopy? A prospective randomized controlled trial. Endoscopy. 2004 Mar;36(3):197-201. doi: 10.1055/s-2004-814247. PMID 14986215
- [Background] Eccleston C, Crombez G. Pain demands attention: a cognitive-affective model of the interruptive function of pain. Psychol Bull. 1999 May;125(3):356-66. doi: 10.1037/0033-2909.125.3.356. PMID 10349356
- [Background] Boselli E. Interest of Analgesia/Nociception Index (ANI) for monitoring the relative parasympathetic tone in anesthetized and awake patients. Douleurs (Paris) (2018)
- [Background] Boselli et al. Analgesia monitoring using Analgesia/Nociception Index: Results of clinical studies in awake and anesthetized patients. Le Praticien en anesthésie réanimation. 2015;19:78-86
- [Background] Logier R, Jeanne M, De Jonckheere J, Dassonneville A, Delecroix M, Tavernier B. PhysioDoloris: a monitoring device for analgesia / nociception balance evaluation using heart rate variability analysis. Annu Int Conf IEEE Eng Med Biol Soc. 2010;2010:1194-7. doi: 10.1109/IEMBS.2010.5625971. PMID 21095676
- [Background] Papaioannou V, Chouvarda I, Gaertner E, Benyamina M, Ferry A, Maurel V, Soussi S, Blet A, Chaouat M, Plaud B, Mebazaa A, Legrand M; PRONOBURN Group. Heart rate variability and cardiac baroreflex inhibition-derived index predicts pain perception in burn patients. Burns. 2016 Nov;42(7):1445-1454. doi: 10.1016/j.burns.2016.04.017. Epub 2016 May 8. PMID 27170468
- [Background] Issa R, Julien M, Decary E, Verdonck O, Fortier LP, Drolet P, Richebe P. Evaluation of the analgesia nociception index (ANI) in healthy awake volunteers. Can J Anaesth. 2017 Aug;64(8):828-835. doi: 10.1007/s12630-017-0887-z. Epub 2017 Apr 21. PMID 28432612
- [Background] Boselli E, Musellec H, Martin L, Bernard F, Fusco N, Guillou N, Hugot P, Paqueron X, Yven T, Virot C. Effects of hypnosis on the relative parasympathetic tone assessed by ANI (Analgesia/Nociception Index) in healthy volunteers: a prospective observational study. J Clin Monit Comput. 2018 Jun;32(3):487-492. doi: 10.1007/s10877-017-0056-5. Epub 2017 Aug 20. PMID 28825157
- [Background] Le Guen M, Jeanne M, Sievert K, Al Moubarik M, Chazot T, Laloe PA, Dreyfus JF, Fischler M. The Analgesia Nociception Index: a pilot study to evaluation of a new pain parameter during labor. Int J Obstet Anesth. 2012 Apr;21(2):146-51. doi: 10.1016/j.ijoa.2012.01.001. Epub 2012 Feb 21. PMID 22360936
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Yi P, Pryzbylkowski P. Opioid Induced Hyperalgesia. Pain Med. 2015 Oct;16 Suppl 1:S32-6. doi: 10.1111/pme.12914. PMID 26461074
- [Background] Maurice-Szamburski A, Loundou A, Capdevila X, Bruder N, Auquier P. Validation of the French version of the Amsterdam preoperative anxiety and information scale (APAIS). Health Qual Life Outcomes. 2013 Oct 7;11:166. doi: 10.1186/1477-7525-11-166. PMID 24099176
- [Background] Facco E, Stellini E, Bacci C, Manani G, Pavan C, Cavallin F, Zanette G. Validation of visual analogue scale for anxiety (VAS-A) in preanesthesia evaluation. Minerva Anestesiol. 2013 Dec;79(12):1389-95. Epub 2013 Jul 9. PMID 23860442
- [Background] Abend R, Dan O, Maoz K, Raz S, Bar-Haim Y. Reliability, validity and sensitivity of a computerized visual analog scale measuring state anxiety. J Behav Ther Exp Psychiatry. 2014 Dec;45(4):447-53. doi: 10.1016/j.jbtep.2014.06.004. Epub 2014 Jun 18. PMID 24978117
- [Background] Hornblow AR, Kidson MA. The visual analogue scale for anxiety: a validation study. Aust N Z J Psychiatry. 1976 Dec;10(4):339-41. doi: 10.3109/00048677609159523. No abstract available. PMID 1071419
- [Background] Kindler CH, Harms C, Amsler F, Ihde-Scholl T, Scheidegger D. The visual analog scale allows effective measurement of preoperative anxiety and detection of patients' anesthetic concerns. Anesth Analg. 2000 Mar;90(3):706-12. doi: 10.1097/00000539-200003000-00036. PMID 10702461
- [Result] Wismeijer AA, Vingerhoets AJ. The use of virtual reality and audiovisual eyeglass systems as adjunct analgesic techniques: a review of the literature. Ann Behav Med. 2005 Dec;30(3):268-78. doi: 10.1207/s15324796abm3003_11. PMID 16336078